CLINICAL TRIAL: NCT05337709
Title: Pharmacist Provided Intervention in Osteoarthritis: Community Pharmacies Based Trial
Brief Title: Pharmacist Provided Intervention (Education and Medication Review) in Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Monash University Malaysia (Other)
Responsible Party: Principal Investigator, Parbati Thapa, PhD Student, Principal Investigator, Monash University Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0
Record Dates: First submitted 2022-04-07; First posted 2022-04-20 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Osteoarthritis; Pain
MeSH Terms: conditions — Osteoarthritis; Pain | interventions — Medication Review

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to either intervention or the control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): Patients from the pharmacies assigned as treatment group will receive intervention. Intervention are education (aid with leaflet and video) and medication review with counselling.
  Interventions: Other: Education intervention and medication review
- control group (No Intervention): Patients from the pharmacies assigned as control group will receive as usual care they have been provided regularly.

INTERVENTIONS:
Other: Education intervention and medication review — Education on osteoarthritis and pain management will be provided to the patients by face-to-face communication at the first meeting, aided with a leaflet, then patients will get the follow-up calls and a video will be shown to enforce the intervention. Medication review includes the assessment of patients' knowledge on the indication, identification of any drug-related problem, and counseling on the proper use of medication.
  Arms: treatment group

SUMMARY:
The purpose of this study is to initiate pharmacist intervention (educational and medication review) among osteoarthritis patients visiting community pharmacies.

DETAILED DESCRIPTION:
Community pharmacists are one of the most accessible health care professionals for patient care in chronic diseases including osteoarthritis and can provide patient education, conduct medication review, and collaborate with the multidisciplinary pain management team, to improve treatment outcomes and quality of life. Studies have reported that pharmacist-provided intervention was beneficial as it increased patients' knowledge of osteoarthritis, reduced the rates of adverse events associated with analgesics, and improved self-perceived health and function. So this study aims to provide intervention through community pharmacists.

Potential patients will be identified from community pharmacies and consent will be obtained from patients before enrolling them in the study. The study will be a cluster-randomized trial. Thus pharmacies will be randomized, either to control or treatment group. Patients in the treatment group will receive the pharmacist-initiated intervention while in the control group will receive usual care.

The intervention will be an education on osteoarthritis, its management, and self-care activities followed by a medication review. Pharmacists assess patients' knowledge of medication indication, identify adverse effects or drug-related problems, and counsel patients on proper medication use.

Education intervention will be provided through face-to-face communication at the time of enrollment and a leaflet will be provided. The patient will receive a phone call and will be able to view the video in the succeeding weeks to enforce the intervention.

Outcome measures will be assessed at baseline, three months, and six months from enrolment in both treatment and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years and above with the complaint of osteoarthritis
* Patient willing to participate in the study
* Patient with chronic pain (persisting for more than three months)

Exclusion Criteria:

* Patient unable to provide the consent due to severe mental health, cognitive impairment or learning difficulties
* Patient with a terminal illness
* Patient having sufficient knowledge on osteoarthritis, its management and self-care activities as assessed from the questionnaire (respond correctly to 80% of the question or above)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline pain intensity at 3 and 6 months | baseline, 3 months and 6 months
  Numeric pain rating scale will be used to measure the pain intensity. The numeric pain rating scale (NPRS) is an 11-point scale. Respondents can choose a number between 0 to 10, where 0 = no pain and 10 = extreme or worst pain. It has shown a high correlation with the visual analogue scale and can be used in rheumatoid arthritis and other types of chronic pain. It can be administered verbally to be done over the telephone. It has been translated into the Nepalese language.
Change from baseline patient's knowledge at 3 and 6 months | baseline, 3 months and 6 months (change in patients knowledge from baseline
  Patient knowledge will be assessed using the questionnaire developed by the principal investigator in consultation with literature review and expert consultation. It consists of 12 questions on osteoarthritis and pain management. It has been translated into Nepalese languages and validated. Correct responses will be counted and presented as percentages. Higher percentages mean better knowledge.
Change from baseline physical function at 3 and 6 months | baseline, 3 months and 6 months
  Western Ontario and Mc Master Universities Arthritis Index (WOMAC) is the tool commonly used for evaluation in osteoarthritis.It consist of 24 items divided into 3 subscales; pain (5 items), stiffness (2 items), physical Function (17 items). Its response is based on a number between 0 to 4, where 0=none, 1=mild, 2=moderate, 3=severe, 4=extreme.

SECONDARY OUTCOMES:
Change from baseline depression score at 6 months | baseline and 6 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) depression scale 8 items: is a set of person-centred measures that evaluates mental health in adults and children. It can be used with the general population and individuals living with chronic conditions. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of depression.
Change from baseline patients quality of life at 6 months | baseline and 6 months
  The quality of life assessment questionnaire EQ-5D-3L (EUROQOL) is one of the most common tools to measure health-related quality of life. It helps to assess the Quality of life-based on five dimensions mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems.
Patient satisfaction | At 6 months of enrollment
  Patient satisfaction will be assessed using the patient satisfaction questionnaire. Higher the score better is the satisfaction level.

CONTACTS AND LOCATIONS:
Locations (1):
- Community Pharmacies, Pokhara, Gandaki, Nepal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McLachlan AJ, Carroll PR, Hunter DJ, Wakefield TAN, Stosic R. Osteoarthritis management: Does the pharmacist play a role in bridging the gap between what patients actually know and what they ought to know? Insights from a national online survey. Health Expect. 2022 Jun;25(3):936-946. doi: 10.1111/hex.13429. Epub 2022 Jan 8. PMID 34997667
- [Background] Kielly J, Davis EM, Marra C. Practice guidelines for pharmacists: The management of osteoarthritis. Can Pharm J (Ott). 2017 May 1;150(3):156-168. doi: 10.1177/1715163517702168. eCollection 2017 May-Jun. No abstract available. PMID 28507652
- [Background] Thapa P, Lee SWH, Kc B, Dujaili JA, Mohamed Ibrahim MI, Gyawali S. Pharmacist-led intervention on chronic pain management: A systematic review and meta-analysis. Br J Clin Pharmacol. 2021 Aug;87(8):3028-3042. doi: 10.1111/bcp.14745. Epub 2021 Feb 24. PMID 33486825
- [Background] Marra CA, Cibere J, Grubisic M, Grindrod KA, Gastonguay L, Thomas JM, Embley P, Colley L, Tsuyuki RT, Khan KM, Esdaile JM. Pharmacist-initiated intervention trial in osteoarthritis: a multidisciplinary intervention for knee osteoarthritis. Arthritis Care Res (Hoboken). 2012 Dec;64(12):1837-45. doi: 10.1002/acr.21763. PMID 22930542
- [Background] Hansson EE, Jonsson-Lundgren M, Ronnheden AM, Sorensson E, Bjarnung A, Dahlberg LE. Effect of an education programme for patients with osteoarthritis in primary care--a randomized controlled trial. BMC Musculoskelet Disord. 2010 Oct 25;11:244. doi: 10.1186/1471-2474-11-244. PMID 20969809
- [Derived] Thapa P, Kc B, Gyawali S, Leong SL, Mohamed Ibrahim MI, Lee SWH. Effectiveness of community pharmacist-led interventions in osteoarthritis pain management: A cluster-randomized trial. Res Social Adm Pharm. 2024 Feb;20(2):149-156. doi: 10.1016/j.sapharm.2023.10.012. Epub 2023 Nov 4. PMID 37945419